CLINICAL TRIAL: NCT02271919
Title: Varenicline and Combined NRT for Initial Smoking Cessation and Rescue Treatment in Smokers: A Randomized Pilot Trial
Brief Title: Varenicline and Combined NRT for Smoking Cessation
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-0213; NCI-2015-00610 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0213 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-10-17; First posted 2014-10-22 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cigarette Smoker; Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Nicotine; Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (varenicline and placebo) (Experimental): Patients receive varenicline orally (PO) once daily (QD) or twice daily (BID), placebo patches QD, and placebo lozenges PO QD beginning on day 9 and continue for 6 weeks. Patients who are abstinent at week 6 will continue treatment for an additional 6 weeks. Patients who fail to achieve abstinence at week 6 are re-randomized to 6 additional weeks of therapy consisting of either continuing on the same treatment, switching to CNRT, or receiving high-dose varenicline. Patients also receive behavioral smoking cessation counseling consisting of 4 in-person visits, 4 phone visits, and 4 brief supportive phone calls lasting 10-15 minutes each over the 12 weeks of treatment.
  Interventions: Drug: Nicotine Lozenge; Drug: Nicotine Patch; Other: Placebo; Other: Tobacco Cessation Counseling; Drug: Varenicline
- Group II (placebo, nicotine patch and lozenge) (Placebo Comparator): Patients receive placebo tablets PO QD or BID, nicotine patches QD, and nicotine lozenges PO QD beginning on day 9 and continue for 6 weeks. Patients who are abstinent at week 6 will continue treatment for an additional 6 weeks. Patients who fail to achieve abstinence at week 6 are re-randomized to 6 additional weeks of therapy consisting of either continuing on the same treatment, switching to varenicline, or receiving high-dose CNRT. Patients also receive behavioral smoking cessation counseling consisting of 4 in-person visits, 4 phone visits, and 4 brief supportive phone calls lasting 10-15 minutes each over the 12 weeks of treatment.
  Interventions: Drug: Nicotine Lozenge; Drug: Nicotine Patch; Other: Placebo; Other: Tobacco Cessation Counseling

INTERVENTIONS:
Drug: Nicotine Lozenge — Given PO
  Other Names: Commit
Drug: Nicotine Patch — Given via patch
  Other Names: NicoDerm CQ; Nicotine Skin Patch; Nicotine Transdermal Patch
Other: Placebo — Given PO or via patch
  Other Names: placebo therapy; PLCB; sham therapy
Other: Tobacco Cessation Counseling — Receive behavioral smoking cessation counseling
Drug: Varenicline — Given PO
  Other Names: Champix; Chantix; CP-526555
  Arms: Group I (varenicline and placebo)

SUMMARY:
This randomized pilot phase IV trial studies the side effects and how well varenicline works compared to nicotine replacement therapy in helping patients that smoke to quit. Varenicline is a drug that acts the same way as nicotine in the brain but is not habit-forming. Nicotine replacement therapy consists of nicotine patches and lozenges. It is not yet known if varenicline is more effective than nicotine replacement therapy in helping patients quit smoking.

DETAILED DESCRIPTION:
Primary Objectives: To estimate (a) the effects at 12 weeks of either continuing on their current medication, switching to the other medication, or increasing the dose of their current medication among smokers initially treated with either varenicline 2 mg (VAR) or nicotine patch + ad lib lozenge (combined nicotine replacement therapy; CNRT) but who relapsed to smoking by week 6 of treatment, and (b) the effects of 12 weeks of continued treatment on either VAR or CNRT among individuals who are abstinent from smoking at 6 weeks.

OUTLINE: Patients are randomized to 1 of 2 groups. GROUP I: Patients receive varenicline orally (PO) once daily (QD) or twice daily (BID), placebo patches QD, and placebo lozenges PO QD beginning on day 9 and continue for 6 weeks. Patients who are abstinent at week 6 will continue treatment for an additional 6 weeks. Patients who fail to achieve abstinence at week 6 are re-randomized to 6 additional weeks of therapy consisting of either continuing on the same treatment, switching to CNRT, or receiving high-dose varenicline. Patients also receive behavioral smoking cessation counseling consisting of 4 in-person visits, 4 phone visits, and 4 brief supportive phone calls lasting 10-15 minutes each over the 12 weeks of treatment.

GROUP II: Patients receive placebo tablets PO QD or BID, nicotine patches QD, and nicotine lozenges PO QD beginning on day 9 and continue for 6 weeks. Patients who are abstinent at week 6 will continue treatment for an additional 6 weeks. Patients who fail to achieve abstinence at week 6 are re-randomized to 6 additional weeks of therapy consisting of either continuing on the same treatment, switching to varenicline, or receiving high-dose CNRT. Patients also receive behavioral smoking cessation counseling consisting of 4 in-person visits, 4 phone visits, and 4 brief supportive phone calls lasting 10-15 minutes each over the 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Smoking 5 or more cigarettes, little cigars and/or cigarillos per day, on average, within the 2 months preceding the screening visit and expired carbon monoxide (CO) greater than or equal to 6 parts per million (ppm) (if less than or equal to 5, then positive cotinine test)
* Interested in treatment that might change smoking behavior
* Able to follow verbal and written instructions in English and complete all aspects of the study
* Provide informed consent and agree to all assessments and study procedures
* Have an address and telephone number where he/she may be reached
* Be the only participant in his/her household

Exclusion Criteria:

* Within the month immediately preceding the screening visit, use of any form of tobacco products other than cigarettes, little cigars and/or cigarillos on 3 or more days within a week if the individual refuses to refrain from such tobacco use during the course of the study
* Current enrollment or plans to enroll in another smoking cessation program in the next 12 months
* Plan to use other nicotine substitutes (i.e., over-the-counter [OTC] or prescription medication for smoking cessation) or smoking cessation treatments in the next 12 months
* Uncontrolled hypertension (systolic blood pressure; [SBP] greater than 180 or diastolic blood pressure; [DBP] greater than 110)
* History of severe kidney disease (e.g. chronic or acute kidney failure) with creatinine clearance below 30 and/or severe liver disease with liver tests over 4 times the upper normal level
* Laboratory evaluations (kidney and liver) outside normal limits and of potential clinical significance in the opinion of the investigator
* Serious or unstable disease within the past 3 months
* History (last 3 months) of abnormal heart rhythms, cardiovascular disease (stroke, angina, heart attack) may result in ineligibility; these conditions will be evaluated on a case by case basis by the study physician
* Current use of certain medications: (1) smoking cessation meds (last 7 days), i.e., Wellbutrin, Bupropion, Zyban, nicotine replacement therapy (NRT), Chantix, (2) certain medications to treat depression (last 14 days), i.e. monoamine oxidase inhibitors (MAOIs) and Elavil (Amitriptyline), (3) a case by case determination will be made by study physician for medication on precautionary list, i.e. nitroglycerin, or (4) daily use of opioids for 30 days or more on phone screen or at screening is exclusionary however pro re nata (PRN) use is allowed (i.e., 3:7 days per week or less or if more frequent, use less than a month's duration)
* Meet criteria for the following psychiatric and/or substance use disorders as assessed by the MINI International Neuropsychiatric Interview (MINI): items C (current manic or hypomanic episode only), I (alcohol abuse - Alcohol Addendum - past 6 months only; current alcohol dependence), J (substance abuse - Substance Abuse Addendum - past 6 months only; current substance dependence), K (current/lifetime psychotic disorder or current/lifetime mood disorder with psychotic features); individuals who meet criteria for non-exclusionary psychiatric disorders that are considered clinically unstable and/or unsuitable to participate as determined by the principal investigator and/or study physician
* Individuals rated as moderate (9-16) to high (17 or greater) on suicidality as assessed by Module B of the MINI
* Psychiatric hospitalization within 1 year of screening date
* A positive urine pregnancy test during the screening period; women who are two years post-menopausal, or who have had a tubal ligation or a partial or full hysterectomy will not be subject to a urine pregnancy test
* Pregnant, breast-feeding or of childbearing potential and is not protected by a medically acceptable, effective method of birth control while enrolled in the study; medically acceptable contraceptives include: (1) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, or (3) an intrauterine device (IUD); contraceptive measures sold for emergency use after unprotected sex are not acceptable methods for routine use
* History of hypersensitivity or allergic reaction to varenicline, NRT, or any component of these formulations
* Any medical or psychiatric condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the principal investigator and/or study physician
* Subject considered by the investigator as unsuitable candidate for receipt of an investigational drug, or unstable to be followed up throughout the entire duration of the study
* Positive toxicology screen for any of the following drugs: cocaine, opiates, methadone, benzodiazepines, barbiturates, amphetamines, methamphetamines, phencyclidine (PCP), or tetrahydrocannabinol (THC); a. participants with valid prescriptions for opiates, benzodiazepines, barbiturates, amphetamines or methadone will not be excluded; b. participants failing the toxicology screen will be allowed to re-screen once; if they test positive again, they will not be allowed to return; study physician may clear participant to continue on if there is a reasonable possibility the positive drug screen is the result of cross-reactivity with the participant's concomitant medications resulting in a false positive

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Seven-day point prevalence and treatment or treatment strategy | At week 6
  Estimated rates of seven-day point prevalence for varenicline and nicotine patch + lozenge at week 6 derive from meta-analyses.
Main effects of varenicline and nicotine patch + lozenge on smokers who remain on these medications throughout the trial as documented in questionnaires | Up to 12 weeks
  Participants complete questionnaires about several topics including depression, mood, smoking behavior, and any effects from the study drug.
Probability of response at week 12 conditional on response at week 6 and continuation of treatment | At 12 weeks
  The probability of response at week 12 conditional on response at week 6 and continuation based on clinical consensus, taking into account the marginal rates of response at twelve weeks reported derived from meta-analysis. Monte Carlo simulations (K = 500) determined predictive power for the planned analyses.
Probability of response at week 12 conditional on non-response at week 6 and continuation of treatment | At 12 weeks
  The probability of response at week 12 conditional on non-response at week 6 and continuation of treatment based on clinical consensus, taking into account the marginal rates of response at twelve weeks reported derived from meta-analysis. Monte Carlo simulations (K = 500) determined predictive power for the planned analyses.
Probability of response at week 12 conditional on non-response at week 6 and augmentation of treatment | At 12 weeks
  The probability of response at week 12 conditional on non-response at week 6 and augmentation of treatment based on clinical consensus, taking into account the marginal rates of response at twelve weeks reported derived from meta-analysis. Monte Carlo simulations (K = 500) determined predictive power for the planned analyses.
Probability of response at week 12 conditional on non-response at week 6 and treatment switching | At 12 weeks
  The probability of response at week 12 conditional on non-response at week 6 and treatment switching based on clinical consensus, taking into account the marginal rates of response at twelve weeks reported derived from meta-analysis. Monte Carlo simulations (K = 500) determined predictive power for the planned analyses.
Probability that treatment continuation, switching, or augmentation confers benefit conditional upon failing to quit after the initial treatment with nicotine patch + lozenge for six weeks | 12 weeks
  Monte Carlo simulations (K = 500) determined predictive power for the planned analyses.
Probability that treatment continuation, switching, or augmentation confers benefit conditional upon failing to quit after initial treatment with varenicline for six weeks | 12 weeks
  Monte Carlo simulations (K = 500) determined predictive power for the planned analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Robinson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Cinciripini PM, Green CE, Shete S, Minnix JA, Robinson JD, Cui Y, Kim S, Kypriotakis G, Beneventi D, Blalock JA, Versace F, Karam-Hage M. Smoking Cessation After Initial Treatment Failure With Varenicline or Nicotine Replacement: A Randomized Clinical Trial. JAMA. 2024 May 28;331(20):1722-1731. doi: 10.1001/jama.2024.4183. PMID 38696203
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT02271919/ICF_000.pdf